CLINICAL TRIAL: NCT00789282
Title: Single-blinded, Two-arm, Randomized Clinical Trial of Patients With Type 2 Diabetes Mellitus That Will Compare'Usual Care' With an 'Enhanced Care' Model of Chronic Disease Management That is Based in the Practices of Family Physicians Participating in Primary Care Networks (PCN's).
Brief Title: Improving the Care of Diabetic Patients: A Randomized Trial of a Family Physician Office-Based Chronic Disease Care Model for Patients With Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges.
Sponsor: University of Alberta (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 200500865; UofA grant #: 20070388
Record Dates: First submitted 2008-05-12; First posted 2008-11-11 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: chronic disease; Family Physician; primary care network; practice-based model; type 2 diabetes; complications; sequelae
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Group (Active Comparator): The 'usual care' study arm (control) will reflect current patterns of care for patients with thpe 2 diabetes in the Capital Health region
  Interventions: Other: reflects current patterns of care
- Enhanced Care Group (Experimental): In the enhanced care group(intervention arm) the participants will receive a multifactorial intervention with three main components that include: optimized medical management, 2) support for development of enhanced patient self management skills, and 3) organized proactive follow-up by chronic disease management teams to support improvement in care.
  Interventions: Other: multidisciplinary approach; Other: multifactorial approach - for enhanced care group

INTERVENTIONS:
Other: multidisciplinary approach — Provides an integrated, proactive approach to the management of patients with chronic diseases (ie: diabetes and sequelae) Wagner Model- care encompassed in 3 overlapping galaxies: wider community; the health care system; and the provider organization. There are 6 essential elements: community resources and policies; health care organization; patient self-management support; delivery system design; decision support; and clinical information systems.
  Arms: Enhanced Care Group
Other: multifactorial approach - for enhanced care group — optimized medical management support for development of enhanced patient self management skills organized proactive follow-up chronic disease management teams
  Arms: Enhanced Care Group
Other: reflects current patterns of care — Continue under the care of their family physician and specialists with referral to diabetic assessment and treatment centers at the discretion of the patient and physician.
  Normal manner of care: could attend diabetic self education classes and consultations regarding management of diabetes. Or, participate in other patient self management program of their choice.
  Arms: Usual Care Group

SUMMARY:
The purpose of the study is to determine the efficacy of a family physician practice-based model of chronic disease management (CDM) based in Primary Care Networks (PCN's) that is integrated with the Capital Health Regional Diabetes Program for care of patients with type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
This is a single-blinded, two-arm, randomized clinical trial of patients with type 2 diabetes mellitus that will compare 'usual care' with an 'enhanced care' model of chronic disease management that is based in the practices of family physicians participating in Primary Care Networks (PCN's).

In this study, patients will be randomized into:

1. Usual care (control) Will reflect current patterns of care for patients with type 2 diabetes in the Capital Health region.
2. Enhanced Care (intervention) Will receive a multifactorial intervention with three main components that include:

   1. optimized medical management,
   2. support for development of enhanced patient self care management skills, and
   3. organized proactive follow-up by chronic disease management (CDM) teams to support improvements in care.

These components are key elements of the Chronic Care Model. They will be delivered by CDM teams working in the practices family physicians in the Primary Care Networks (PCN's).

Clinical Outcome Measures

* will be assessed at baseline, 3 months, and 6 months.

Quality of Life Measures

* will be measured at baseline, 6 months, and 12 months.

Risks and Benefits

The prevalence of diabetes mellitus is high and expected to increase in the future. It is unlikely that current systems of care will be adequate to provide care to patients with diabetes in the future. This study will evaluate a model of care of care , based on the Chronic Care Model, which has been provided to improve the care of patients with chronic diseases like diabetes. Patients may benefit due to improved care for their diabetes. Health care providers may benefit through an increased understanding of best methods and organization to provide care to populations of patients with diabetes and other chronic diseases.

Privacy and Confidentiality:

All study data collected will be kept confidential. Respondents will not be identified by name in any presentation or publications arising from the study. Access to data is restricted to investigators and project staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes (2003 classification by the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus) receiving any therapy with HbA1c of > or = 7.0% between the ages of 40 - 75 years.

Exclusion Criteria:

* Type 1 diabetes
* Pregnancy
* Severe diabetic complications that include end stage renal disease requiring dialysis
* Proliferative retinopathy (growth of new vessels on the retina and posterior surface of the vitreous that requires laser therapy)
* Uncontrolled cardiovascular disease (CVS event within 1 year of enrollment)
* Psychiatric disease or cognitive impairment that would interfere with treatment compliance
* Cancer or terminally ill patients with less than 6 months life expectancy
* Blindness
* Other severe co- morbid diseases
* Participation in another intense multifactorial intervention for the management of type 2 diabetes
* Participation in another study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
A higher proportion of patients with type 2 diabetes enrolled in the 'enhanced care' arm compared with the patients enrolled 'usual' care' arm will achieve an absolute reduction in their HbaA1c of 1.0% or greater during the study period. | 1 year

SECONDARY OUTCOMES:
A higher proportion of patients with type 2 diabetes in the 'enhanced care' arm compared with the patients enrolled in 'usual care' arm will achieve a 10% or greater reduction in HbA1c values during the study period. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bell, MD,MSc,CCFP,FCFP, Principal Investigator — Professor, Dept of Family Medicine, University of Alberta
Locations (1):
- University of Alberta, Dept of Family Medicicne, Edmonton, Alberta, Canada